CLINICAL TRIAL: NCT06142695
Title: Ultrasonic Evaluation of Carbon Dioxide Laser Effects on Patients With Genitourinary Syndrome
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, VILLA PAOLA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4689
Record Dates: First submitted 2023-07-18; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Genitourinary Syndrome of Menopause

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study was to evaluate the efficacy of vaginal Carbon Dioxide Laser treatment in patients with Genitourinary Syndrome of Menopause on the improvement of Vulvovaginal Atrophy (VVA) and stress urinary incontinence (SUI) by objective parameters and in particular to assess the ultrasound measurement of specific vaginal parameters in order to evaluate a new objective tool of assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age <75 years, menopause (naturally, pharmacologically or surgically induced, at least 12 months)
* Negative Papanicolaou test (PAP) performed within 12 months before enrolment. and one of the following:
* Presence of vulvovaginal atrophy [vaginal health index (VHI) < 15]
* Initial Urinary Incontinence based on patient history = 1 (according to the "Stamey incontinence score of Stress Urinary Incontinence" - min. 0 = no incontinence, max. 3 = severe incontinence)
* Standardized stress provocation test

Exclusion Criteria:

* Age >45 years
* The presence of vaginal lesions (active or in the previous 30 days).
* genitourinary tract infection.
* abnormal uterine bleeding.
* use of hormone replacement therapy up to 6 months before enrolment.
* history of photosensitivity disorder or use of photosensitizing drugs.
* genitals prolapse (grade II - III according to the Pelvic Organ Prolapse Quantification)
* a serious or chronic condition that could interfere with study compliance.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Menopausal patients that attended our clinic of menopausal disorders and performed Carbon Dioxide Laser therapy for genitourinary syndrome.
  In order to enroll patients with Genitourinary Syndrome of Menopause, the investigator used the Vaginal Health Index (VHI), Vulvar Health Index (VuHI), and Stress Urinary Incontinence (SUI) scales.
  * The VHI score assesses vaginal health, with a cutoff of <15 on the index to diagnose patients with atrophy [ranging from "complete atrophy" (0) to "optimal vaginal health" (25)].
  * The VuHI score assesses vulvar health, on a scale from normal (0) to severe (3). The overall score ranges from 0 to 24, and its cutoff for diagnosing atrophic vulva is >8 on the index.
  * Stress Urinary Incontinence (SUI) is characterized by sudden urine loss. Evaluated using the Stamey score, with ratings of no incontinence (0) to severe incontinence (3).
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2022-01-09 (Actual)

PRIMARY OUTCOMES:
Evaluating the effectiveness of Carbon Dioxide Laser in patients with genitourinary syndrome of menopause in terms of the improvement in a specific vaginal ultrasonographic parameters | 4 months
  To evaluate the primary outcome, we examined the following vaginal ultrasonographic parameters (by transvaginal probe), both before and after 3 vaginal Carbon Dioxide Laser applications:
  * Thickness of the anterior vaginal walls (VWT) at the level of the introitus of the inferior vaginal third (expressed in millimeters);
  * Thickness of the posterior VWT at the level of the introitus of the inferior vaginal third (expressed in millimeters).
  Positive outcomes are evidenced if thickness (expressed in millimeters) is increased after treatment in both anterior and posterior vaginal walls.

CONTACTS AND LOCATIONS:
Locations (1):
- FPG gemelli RCCS, Rome, Lazio, Italy